CLINICAL TRIAL: NCT05761093
Title: A Study to Evaluate Patient and Physician Benefit/ Risk Preferences for Treatment of Metastatic Prostate Cancer (mPC) in Hong Kong: a Discrete Choice Experiment
Brief Title: Patient and Physician Benefit/ Risk Preferences for Treatment of mPC in Hong Kong: a Discrete Choice Experiment
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, NG Chi Fai, Professor, Chinese University of Hong Kong
Other Study IDs: CRE-2022.301
Record Dates: First submitted 2023-02-28; First posted 2023-03-09 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to examine the preference weightings in term of risk/ benefit attributes of treatment in physician and prostate cancer patients from different stages of disease.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older,
* diagnosis of metastatic prostate cancer within 5 years,
* able to read and write,
* accepting and signing the informed consent

Exclusion Criteria:

* if patients are unable to complete the survey by themselves due to physical or psychological reasons,
* deemed ineligible by treating physicians if patients are unable to complete the survey by themselves due to physical or psychological reasons,
* deemed ineligible by treating physicians

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: 300 consecutive patients with metastatic prostate cancer (150 mHSPC and 150 mCRPC) within 5 years will be recruited
Sampling Method: Non-Probability Sample
Enrollment: 306 (Estimated)
Dates: Start 2022-09-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Patient preferences for treatment attributes in prostate cancer from different stages of disease | 15 minutes (Once through survey)
  Derived from discrete choice experiment
The Preference weighting from Physicians involved in the treatment of prostate cancer in term of risk/benefit attributes of treatment. | 15 minutes (Once through survey)
  Derived from discrete choice experiment.

SECONDARY OUTCOMES:
To examine the effect of socio-economic status on preference weighing | 15 minutes (Once through survey)
  Derived from discrete choice experiment
To examine the status of comorbidities on preference weighing | 15 minutes (Once through survey)
  Derived from discrete choice experiment
To examine their willingness of trading off survival with improving QOL | 15 minutes (Once through survey
  Derived from discrete choice experiment

CONTACTS AND LOCATIONS:
Overall Officials: Chi Fai NG, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sartor O, de Bono JS. Metastatic Prostate Cancer. N Engl J Med. 2018 Feb 15;378(7):645-657. doi: 10.1056/NEJMra1701695. Epub 2018 Feb 7. No abstract available. PMID 29412780
- [Background] Feldman-Stewart D, Brundage MD, Van Manen L, Svenson O. Patient-focussed decision-making in early-stage prostate cancer: insights from a cognitively based decision aid. Health Expect. 2004 Jun;7(2):126-41. doi: 10.1111/j.1369-7625.2004.00271.x. PMID 15117387
- [Background] Aning JJ, Wassersug RJ, Goldenberg SL. Patient preference and the impact of decision-making aids on prostate cancer treatment choices and post-intervention regret. Curr Oncol. 2012 Dec;19(Suppl 3):S37-44. doi: 10.3747/co.19.1287. PMID 23355792
- [Background] Uemura H, Matsubara N, Kimura G, Yamaguchi A, Ledesma DA, DiBonaventura M, Mohamed AF, Basurto E, McKinnon I, Wang E, Concialdi K, Narimatsu A, Aitoku Y. Patient preferences for treatment of castration-resistant prostate cancer in Japan: a discrete-choice experiment. BMC Urol. 2016 Nov 4;16(1):63. doi: 10.1186/s12894-016-0182-2. PMID 27814714
- [Background] Hauber AB, Arellano J, Qian Y, Gonzalez JM, Posner JD, Mohamed AF, Gatta F, Tombal B, Body JJ. Patient preferences for treatments to delay bone metastases. Prostate. 2014 Nov;74(15):1488-97. doi: 10.1002/pros.22865. Epub 2014 Aug 17. PMID 25132622
- [Background] Ryan M, Farrar S. Using conjoint analysis to elicit preferences for health care. BMJ. 2000 Jun 3;320(7248):1530-3. doi: 10.1136/bmj.320.7248.1530. No abstract available. PMID 10834905
- [Background] Fizazi K, Shore N, Tammela TL, Ulys A, Vjaters E, Polyakov S, Jievaltas M, Luz M, Alekseev B, Kuss I, Kappeler C, Snapir A, Sarapohja T, Smith MR; ARAMIS Investigators. Darolutamide in Nonmetastatic, Castration-Resistant Prostate Cancer. N Engl J Med. 2019 Mar 28;380(13):1235-1246. doi: 10.1056/NEJMoa1815671. Epub 2019 Feb 14. PMID 30763142
- [Background] Gravis G, Fizazi K, Joly F, Oudard S, Priou F, Esterni B, Latorzeff I, Delva R, Krakowski I, Laguerre B, Rolland F, Theodore C, Deplanque G, Ferrero JM, Pouessel D, Mourey L, Beuzeboc P, Zanetta S, Habibian M, Berdah JF, Dauba J, Baciuchka M, Platini C, Linassier C, Labourey JL, Machiels JP, El Kouri C, Ravaud A, Suc E, Eymard JC, Hasbini A, Bousquet G, Soulie M. Androgen-deprivation therapy alone or with docetaxel in non-castrate metastatic prostate cancer (GETUG-AFU 15): a randomised, open-label, phase 3 trial. Lancet Oncol. 2013 Feb;14(2):149-58. doi: 10.1016/S1470-2045(12)70560-0. Epub 2013 Jan 8. PMID 23306100